CLINICAL TRIAL: NCT05592964
Title: The Effect of Oral Fluid Administration 1 Hour Before Surgery on Preoperative Anxiety and Gastric Volume in Pediatric Patients
Brief Title: The Effect of Oral Fluid Administration 1 Hour Before Surgery on Preoperative Anxiety and Gastric Volume in Pediatrics
Status: Completed | Type: Observational
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Zehra Hatipoglu, MD, associate professor, Cukurova University
Other Study IDs: 10/2022
Record Dates: First submitted 2022-10-05; First posted 2022-10-25 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Preoperative Anxiety
Keywords: preoperative period; carbohydrate; anxiety; ultrasonography; pediatrics
MeSH Terms: conditions — Anxiety Disorders | interventions — Angptl4 protein, mouse; Water

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A: Standard fasting group.
  Interventions: Dietary Supplement: Fasting
- Group S: The patient group who were given oral 5 ml/kg (maximum 250 ml) of water 1 hour ago.
  Interventions: Dietary Supplement: Water
- Group K: The patient group who were given an oral 5 ml/kg (maximum 250 ml) carbohydrate rich clear liquid 1 hour ago.
  Interventions: Dietary Supplement: Carbohydrate fluid

INTERVENTIONS:
Dietary Supplement: Fasting — Standard fasting
  Groups: Group A
Dietary Supplement: Water — In Group S, water was given 1 hour before the operation.
  Groups: Group S
Dietary Supplement: Carbohydrate fluid — In Group K, carbohydrate fluid was given 1 hour before the operation.
  Groups: Group K

SUMMARY:
It is a randomized, controlled and prospectively planned observational study.In our study, oral fluid administration 1 hour before surgery in children aged 5-12 years was aimed at preoperative anxiety level as the primary objective; The secondary objective is to evaluate the effects on gastric volume, hemodynamics and blood sugar.The study included 90 paediatric patients aged 5-12 years with ASA score 1-2. Group A (n=30): Standard fasting group. Group S (n=30): A group of patients who were given oral 5 ml/kg (maximum 250 ml) of water 1 hour ago. Group K (n=30): A group of patients who were given an oral 5 ml/kg (maximum 250 ml) carbohydrate rich clear liquid 1 hour ago. All patients were evaluated with the modified Yale Preoperative Anxiety Scale (m-YPAS) before and 1 hour after fluids were administered. After anesthesia, gastric antrum cross-sectional area (GACSA) was measured. Gastric residual volume (GRV) values were calculated. Hemodynamic data, blood sugar levels and parental satisfaction were recorded.

DETAILED DESCRIPTION:
The study included 90 patients between the ages of 5 and 12 with an ASA Score of 1-2 who were scheduled for elective surgery (circumcision, strabismus, orchiopexy, hypospadias, splenectomy, vaginoplasty, laparoscopic gonadal research, epididymis cyst, inguinal hernia). ASA 3-4 was planned to exclude patients with a functional or anatomical disease related to the gastrointestinal tract, those with severe liver, kidney, cardiac or neurological disease, patients using proton pump inhibitor or histamine 2 receptor blocker. Parents and children were informed about the study during the preoperative visit; written and verbal consents were obtained from those who accepted. Patients who participated in the study were randomly divided into three groups:Group A (n=30): Standard fasting group. Group S (n=30): A group of patients who were given oral 5 ml/kg (maximum 250 ml) of water 1 hour ago. Group K (n=30): A group of patients who were given an oral 5 ml/kg (maximum 250 ml) carbohydrate rich clear liquid 1 hour ago.Demographic data (gender, age, height, weight, body mass index (BMI), ASA score and co-morbidity) of the children taken to the preoperative waiting room were recorded. None of them underwent premedication. Patients in all groups were evaluated with m-YPAS score (basal). Patients in Group S and K were then given oral fluid; similarly, after 1 hour, patients in all groups were again evaluated with m-YPAS score.Standard monitoring (electrocardiography, peripheral oxygen saturation and noninvasive blood pressure) was applied to all patients who were taken to the operating room with their parents 1 hour after oral fluids were administered. After the induction of anesthesia was achieved with 2 mg/kg propofol (iv) and 0.6 mg/kg rocuronium (iv), intubation was performed with endotracheal tube appropriate for the age of the children. Anesthesia maintenance was achieved with 2% sevofluran and N2O/O2 40/60% inhalation anesthetics. Ringer Lactate 5-10 ml/kg was preferred for intravenous fluid maintenance.Patients were given the right lateral decubitus position after intubation. GACSA was identified by convex ultrasound (Esaote, myLabtm Six) probe in the abdominal setting, left lobe of the liver and superior mesenteric vein in the sagittal plane. GACSA was measured by determining the anterior-posterior (D1) and cranial-caudal (D2) distances (GAA: D1 x D2 x π / 4). The volume of gastric residue was calculated using a mathematical formula [GRV:-7.8 + (3.5xGAA) + 0.127xage (monthly)]. .In the study, there were two different people who evaluated the basal and m-YPAS scores 1 hour later and performed abdominal USG and were blind.Complications such as vomiting and aspiration that may occur during induction of anesthesia were recorded. Glucose measurement with glucometer (Freestyle Optimum Neo H) was performed at the 20th minute. Systolic blood pressure (SBP), diastolic blood pressure (DBP), mean arterial pressure (OAB), heart rate (HR) were recorded before induction and at intervals of 5 minutes for the first 20 minutes after induction.At the end of surgery, a combination of 0.015 mg/kg atropine + 0.05 mg/kg neostigmine (iv) was applied to terminate the neuromuscular block. After it was decided that breathing and muscle activity were at an adequate level, tracheal extubation was performed and the patient was taken to the recovery room. Parental satisfaction (very good, good or dissatisfied) was assessed in the recovery room. According to the modified Aldrete compilation scoring, patients who scored 9 ≥ were sent to the their bed.

ELIGIBILITY:
Inclusion Criteria:

* ages of 5 and 12
* ASA Score of 1-2

Exclusion Criteria:

* ASA 3-4
* functional or anatomical disease related to the gastrointestinal tract, those with severe liver, kidney, cardiac or neurological disease
* patients using proton pump inhibitor or histamine 2 receptor blocker.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: It was carried out by the Pediatric Surgery and Eye Departments in children who underwent elective surgery.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2022-03-04 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of the Preoperative anxiety scores | Change from Baseline modified yale preoperative anxiety scale 1 hour after fluid
  Modified Yale Preoperative Anxiety Scale (Scores: minimum:23.3-maximum:100) All children were evaluated with mYPAS (basal) when they came to the preoperative preparation room. Group S and K were then given oral fluid; similarly, after 1 hour, patients in all groups were again evaluated with m-YPAS score.
  The mYPAS is performed in children aged 5 to12 years old, both in the preoperative unit and during anesthesia induction, and it is widely used to evaluate children's anxiety before surgery, at the present time

SECONDARY OUTCOMES:
Evaluation of the Gastric residual volume values | after 10 minutes anesthesia induction
  Measurement of gastric sections under ultrasound guidance. After intubation, gastric antral cross-sectional area was measured by ultrasound. Gastric residual volume (GRV) values were calculated.
Evaluation of the blood pressures | Change from SBP, DBP, and MAP at 20 minutes.
  noninvasive blood pressure measurement Systolic blood pressure (SBp), diastolic blood pressure (DBP), mean arterial pressure (MAP) were recorded before induction and at 5-minute intervals for the first 20 minutes after induction.
Blood sugar | at the 20th minute.
  Glucose measurement with glucometer
Evaluation of heart rates | Change from heart rates at 20 minutes.
  Heart rates were recorded before induction and at 5-minute intervals for the first 20 minutes after induction.

CONTACTS AND LOCATIONS:
Locations (1):
- Cukurova University, Faculty of Medicine, Department of Anesthesiology and Reanimation, Adana, Saricam, Turkey (Türkiye)